CLINICAL TRIAL: NCT06521593
Title: Tourniquet in Total Knee Replacement Short and Long Duration: A Comparative Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-414-2021
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Tourniquet Palsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: patients were in the operation room and werent aware of
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients who underwent short duration applying of tourniquet. (Active Comparator): All patients underwent spinal anesthesia and the tourniquet was applied to the middle of the thigh; in group one who underwent long-duration application of a tourniquet, it was applied only before the skin incision by inflating it to 150 mmHg above the systolic blood pressure of the patients and deflation just before cementing
  Interventions: Procedure: Applying a tourniquet for either a short or long time during total knee replacement
- patients who underwent long duration applying of tourniquet. (Experimental): All patients underwent spinal anesthesia and the tourniquet was applied to the middle of the thigh; in group one who underwent long-duration application of a tourniquet, it was applied only before the skin incision by inflating it to 150 mmHg above the systolic blood pressure of the patients and deflation finishing of bone cementation
  Interventions: Procedure: Applying a tourniquet for either a short or long time during total knee replacement

INTERVENTIONS:
Procedure: Applying a tourniquet for either a short or long time during total knee replacement — All patients underwent spinal anesthesia and the tourniquet was applied to the middle of the thigh; in group one who underwent long-duration application of a tourniquet, it was applied only before the skin incision by inflating it to 150 mmHg above the systolic blood pressure of the patients and deflation finishing of bone cementation while in group two who underwent short duration application of a tourniquet, the tourniquet was only applied just before cementation, was inflated also to 150 mmHg above the systolic blood pressure of the patients, and was deflated after bone cementation.

SUMMARY:
Total knee arthroplasty (TKA) is an effective treatment in severe osteoarthritis. We aim to compare the advantages and disadvantages related to the duration of tourniquet application in TKA surgeries.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is considered an effective method in relieving pain and regaining function in severe osteoarthritis patients; however, it is associated with increased blood loss risk which can increase the need for blood transfusion. Tourniquet use during surgery is controversial as it provides a clear visualization which decreases the blood loss and ensures proper cementation which makes it used frequently during TKA. However, its use is associated with complications like nerve palsy, thigh pain, swelling, joint stiffness, wound complications, subcutaneous fat necrosis, vascular injury, deep venous thrombosis (DVT), and prolonged duration of quadriceps recovery.

The proper duration of tourniquet application is also controversial as it affects TKA postoperative outcomes as increasing tourniquet application duration can aggravate the complications risk because of the increased tissue exposure to ischemia. Therefore, minimization of the tourniquet application duration is important which makes researchers investigate if tourniquet application during the cementation process only in TKA could decrease the complications and fasten the recovery.

Limited tourniquet application during TKA decreased swelling and joint pain while it was not associated with blood loss, recovery, or operation time. While applying a tourniquet only in cementation could reduce blood loss, fasten the recovery period, and reduce pain after TKA surgery.

However, decreasing tourniquet application to be only during cementation was associated with increased blood transfusion risk which indicated that this approach was impractical if there was not any improvement in recovery. Therefore, a balance should exist between the increased blood loss and blood transfusion risk during cementation tourniquet application. Therefore, the application time of a tourniquet during cementation in TKA is controversial and no meta-analysis compared using a tourniquet only to the long tourniquet use in TKA surgeries.

Therefore, randomized controlled trials (RCTs) are needed to compare which strategy is better which made us perform this study to compare both strategies regarding pain, Oxford Knee Score (OKS), hospital stay, pain, Knee Society Score (KSS), blood loss, and range of motion (ROM).

ELIGIBILITY:
Inclusion Criteria:

* We included symptomatic grade IV knee primary osteoarthritis cases who were candidates for TKA surgery

Exclusion Criteria:

* we excluded patients with a history of post-infection or traumatic osteoarthritis, knee deformity, hematological diseases, currant infection focus, immune-suppression, or inflammatory arthritis.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss | immediately post operative
  We measured the intraoperative blood loss by subtracting saline volume used in washing from the whole suction volume which was added to the value resulting from subtracting dry foments weight from the wet foments weight used in managing bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
May be shared upon reasonable request